CLINICAL TRIAL: NCT02239341
Title: Effects of Two In-hospital Antepartum Interventions on Functional Ability and Quality of Life in Early Postpartum Women.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Michelle Mottola, Dr., University of Western Ontario, Canada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 105699
Record Dates: First submitted 2014-09-08; First posted 2014-09-12 (Estimated); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: High-Risk Pregnancy
Keywords: hospitalized; activity restriction; bed rest; antepartum; pregnant; high risk

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Music Intervention (M) (Active Comparator): The M intervention will be 30 minutes (same amount of time as E group), but the participants will simply be listening to the same music in bed with no exercise component. They will be wearing the heart rate monitor as in the E group. The M group will act as a control group for the E group.
  Interventions: Other: Music Intervention
- Muscle Conditioning Intervention (E) (Experimental): E (exercise) is 30 minutes in length and will consist of 5 minutes of warm-up, 20 minutes of light strengthening exercises using a theraband, and 5 minutes of cool-down. All exercises will be completed in bed. Each participant will be listening to the same music (as the M group) during exercise. A heart rate monitor will be worn throughout each session. The first session for each participant will be used to complete baseline measurements and to assess initial muscle strength. Difficulty level will be adjusted by using different strength therabands.
  Interventions: Other: Music Intervention; Other: Muscle Conditioning Intervention

INTERVENTIONS:
Other: Music Intervention — Music will be about 120 beats per minute and the participants will listen to the music while wearing head-phones in bed.
Other: Muscle Conditioning Intervention — Music will be about 120 beats per minute and the participants will listen to the music while wearing head-phones and also participate in the muscle conditioning program while in bed.
  Arms: Muscle Conditioning Intervention (E)

SUMMARY:
The current standard of care for pregnant women deemed to be high-risk often involves recommending varying levels of activity-restriction, up to and including hospitalization. High levels of activity-restriction can lead to physical deconditioning of the mother, which can be difficult to recover from after birth. The proposed study will investigate whether a mild muscular conditioning program conducted in bed and given to hospitalized activity-restricted high-risk pregnant women will improve functional ability, cardiovascular deconditioning and overall quality of life in the postpartum period compared to a control group with no in hospital bed-rest exercise program. We hypothesize that women with a in-hospital muscle conditioning program will be better able to perform functional ability tasks and activities of daily living than a control group with no exercise program.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized high-risk pregnant women in hospital for at least 7 days
* Diagnosed with gestational hypertension
* Diagnosed with preeclampsia (mild to moderate)
* Diagnosed with intrauterine growth restriction
* Single baby
* Expecting twins
* Expecting triplets
* Diagnosed with shortened cervix
* Diagnosed with threatened pre-term labour (not actively contracting)

Exclusion Criteria:

* Diagnosed with symptomatic placenta previa (bleeding)
* Diagnosed with severe pre-eclampsia (immediate delivery)
* Diagnosed with conditions indicating a short term hospital stays of less than 7 days
* Diagnosed with infections
* Diagnosed with heart and renal disease
* Diagnosed with diabetes
* Diagnosed with metabolic bone disease
* Diagnosed with hyper-or-hypo-thyroidism
* Diagnosed with Cushing disease and anemia
* Women carrying more than 3 babies

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-10-30 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
Score on the Functional Mobility Assessment Tool | 2 weeks post delivery
  The Functional Mobility Assessment Tool was adapted from a senior fitness test, which uses 7 tests to assess muscular strength, aerobic endurance, flexibility and agility (Chair Stand Test, Arm Curl Test, 6-Minute Walk Test, 2-Minute Step Test, Chair Sit-And-Reach Test, Back Scratch Test, and 8-Foot-Up-And-Go Test).

SECONDARY OUTCOMES:
Quality of life | Baseline (> 28 weeks gestation); 2 weeks post delivery; 2, 6 and 12 months post delivery
  The secondary outcome of the study is to examine quality of life in the postpartum period. Quality of life will be measured by completing four surveys the EQ-5D, and the Postpartum Psychological Profile Questionnaire which includes the Depression Scale (1 page), the State Anxiety Index (1 page) and the Postpartum Physical and Psychological Symptoms Report .
Follow up to Primary outcome Score for Functional Mobility Assessment Tool | 2, 6 and 12 months
  Changes over time within groups and between groups in the post partum period

CONTACTS AND LOCATIONS:
Overall Officials: Michelle F Mottola, PhD, Principal Investigator — University of Western Ontario, Canada
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada